CLINICAL TRIAL: NCT02978105
Title: Effects of Self-conditioning Techniques in Promoting Weight Loss in Patients With Severe Obesity. A Randomized Controlled Trial
Brief Title: Effects of Self-conditioning Techniques in Promoting Weight Loss in Patients With Obesity. A Randomized Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Simona Bo, Associate Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sbo2015
Record Dates: First submitted 2016-11-26; First posted 2016-11-30 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Standard of Care; Diet; Exercise; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): self-conditioning techniques plus standard care
  Interventions: Other: self-conditioning techniques; Other: standard care (diet, exercise and behavioral therapy)
- Control (Active Comparator): Standard care: dietary recommendations, exercise recommendations, and behavioral recommendations
  Interventions: Other: standard care (diet, exercise and behavioral therapy)

INTERVENTIONS:
Other: self-conditioning techniques — Self-hypnosis to increase self-control before meals and every food compulsion episode
  Arms: Experimental
Other: standard care (diet, exercise and behavioral therapy) — dietary recommendations, exercise recommendations, and behavioral recommendations

SUMMARY:
The investigators hypothesized that hypnosis is an alternative technique that could be applied to help patients with obesity to lose weight.

The possibility that a self-conditioning technique (self-hypnosis) added to traditional approach (diet, exercise and behavioral recommendations) will be effective in determining weight loss with respect to the traditional approach in subjects with a body mass index (BMI) between 35 and 50 kg/m2 will be studied.

DETAILED DESCRIPTION:
Obesity is a serious health concern. Most lifestyle interventions fail over time; indeed, overeating often involves loss of control and compulsive behaviors.

Hypnosis could increase the ability to control emotional impulses. Self-conditioning techniques borrowed from hypnosis (self-hypnosis) increase self-control and self-management of emotions. Recent hypnosis techniques with a rapid-induction phase allow the trained patients to go into self-hypnosis in a few minutes and to repeat the experience in complete autonomy, employing a short time of the day only.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent
* BMI between 35 and 50 kg/m2
* Age 20-70 years

Exclusion Criteria:

* Current or previous mental disorders and/or on any psychotropic drug
* Insulin treatment
* Candidates for bariatric surgery
* Current (or discontinued for less than 6 months) treatment with anti-obesity drugs
* Patients at risk of heart failure, edema, ascites (heart diseases, chronic liver diseases, nephrotic syndrome, renal failure)
* Patients with untreated or uncompensated thyroid diseases

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
weight loss | 12 months after randomization

SECONDARY OUTCOMES:
Change in body fat percentage | 12 months after randomization
  Dual Energy X-Ray Absorptiometry (DEXA)
Change in fasting glucose | 12 months after randomization
Change in insulin circulating values | 12 months after randomization
Change in quality of life | 12 months after randomization
  EuroQol (EQ)-5D [Index and Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Simona Bo, MD, Principal Investigator — University of Turin, Italy
Locations (1):
- Città della Salute e della Scienza di Torino, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bo S, Rahimi F, Goitre I, Properzi B, Ponzo V, Regaldo G, Boschetti S, Fadda M, Ciccone G, Abbate Daga G, Mengozzi G, Evangelista A, De Francesco A, Belcastro S, Broglio F. Effects of Self-Conditioning Techniques (Self-Hypnosis) in Promoting Weight Loss in Patients with Severe Obesity: A Randomized Controlled Trial. Obesity (Silver Spring). 2018 Sep;26(9):1422-1429. doi: 10.1002/oby.22262. PMID 30226009